CLINICAL TRIAL: NCT06497803
Title: The Effect of Nurse-Led Body Protection Education on the Sexual Abuse Knowledge Levels of Students With Visual Impairments: A Randomized Controlled Trial
Brief Title: The Effect of Nurse-Led Body Protection Education in Students With Visual Impairments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09.2020.172
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Child Sexual Abuse; Disability, Vision
Keywords: Child sexual abuse; Visually impaired children; Prevention; Health education; Public health nursing
MeSH Terms: conditions — Vision Disorders; Health Education

STUDY DESIGN:
Intervention Model Description: This study is parallel group randomized controlled study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Nurse-led body protection education was provided to the intervention group in groups of 3-4 in 40 minutes. The education was provided as verbal narration by using a doll and distress whistle. In addition, two weeks after the post-test, a reminder education brochure prepared with the braille alphabet was distributed to the students in the intervention group.
  Interventions: Other: Nurse-Led Body Protection Education; Other: Reminder Education Brochure
- Control Group (No Intervention): Pretest, posttest and follow-up test were applied simultaneously to the intervention group and the control group. Throughout the research, the control group continued their routine education. After the follow-up test, the control group was also provided with nurse-led body protection education.

INTERVENTIONS:
Other: Nurse-Led Body Protection Education — Based on BST and Safe Touches education programs and in line with the studies conducted in the literature on children who are not visually impaired, NLBPE was created by the researchers (Akgul et al., 2021; Citak-Tunc et al., 2018; Pulido, 2019; Wurtele, 2007). The program aims to teach visually impaired children how to protect the private parts of their bodies, to distinguish between good and bad touch, to distinguish between good and bad secrets, to say no, scream, and ask for help when necessary. As education tools, dolls and distress whistles were used. In order for children to learn the private parts of their bodies, a doll was used. The practice of "Say No, Scream, Run, and Blow Your Whistle While Running" in order for the students to protect their body from bad touch was applied by the students one by one firstly, and in groups later.
  Other Names: NLBPE
  Arms: Intervention Group
Other: Reminder Education Brochure — The brochure was prepared in line with the NLBPE and included what is a good touch and a bad touch, how to distinguish a good touch from a bad touch, examples of good touch and bad touch, and what to do when encountered with a bad touch (Say No, Scream, Run, and Blow Your Whistle While Running). The brochure, the content of which was prepared by the researcher, was translated into Braille Alphabet by a visually impaired teacher working at the school where the research was conducted, before it was distributed to the intervention group members.
  Other Names: REB
  Arms: Intervention Group

SUMMARY:
In the study, it was aimed to examine the effect of nurse-led body protection education on the sexual abuse knowledge levels of students with visual impairments.

DETAILED DESCRIPTION:
Children with visual impairments form a risky group in terms of abuse as they are more dependent in relation to providing self-care compared to children with visually healthy and they use their sense of touch in communicating with the environment. The 53 students with visual impairments were randomly assigned to the intervention group and the control group. The study data were collected through children's knowledge of abuse questionnaire - revised with the subdimensions of good touch and bad touch. Nurse-led body protection education was provided to the intervention group in groups of 3-4 in 40 minutes. The education was provided as verbal narration by using a doll and distress whistle. In addition, two weeks after the post-test, a reminder education brochure prepared with the braille alphabet was distributed to the students in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Students with visual impairments who gave their consent to participate in the study and who could communicate in Turkish were included in the study.

Exclusion Criteria:

* Students who had a mental disability in addition to visual impairment were excluded from the study.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
The Good Touch subscale of the Children's Knowledge of Abuse Questionnaire-Revised scale | Change in knowledge level within two months
  The Good Touch subscale of the Children's Knowledge of Abuse Questionnaire-Revised scale was applied in the pre-test, post-test and follow-up test. The scale was developed by Tutty in 1992 and finalized by revising in 1995 (Tutty, 1997). The Turkish adaptation study of the scale was conducted by Yilmaz and Cenkseven-Onder (2020). Eight items on the scale (1, 3, 8, 17, 20, 25, 27 and 30) are under the Good Touch subdimension. The responses to the items are in the form of Correct, Incorrect, and Don't Know. In the analysis of the scale, "correct" answers are scored as 1 point, and "incorrect" and "Don't Know" responses are scored as 0 point.
The Bad Touch subscale of the Children's Knowledge of Abuse Questionnaire-Revised scale | Change in knowledge level within two months
  The Bad Touch subscale of the Children's Knowledge of Abuse Questionnaire-Revised scale was applied in the pre-test, post-test and follow-up test. The scale was developed by Tutty in 1992 and finalized by revising in 1995 (Tutty, 1997). The Turkish adaptation study of the scale was conducted by Yilmaz and Cenkseven-Onder (2020). 22 items are under the Bad Touch subdimension. The responses to the items are in the form of Correct, Incorrect, and Don't Know. In the analysis of the scale, "correct" answers are scored as 1 point, and "incorrect" and "Don't Know" responses are scored as 0 point.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Ergun, Prof, Study Chair — Marmara University; Esma Akgul, MSc, RN, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cecen-Erogul AR, Kaf Hasirci O. The effectiveness of psycho-educational school-based child sexual abuse prevention training program on turkish elementary students. Educational Sciences: Theory and Practice. 2013; 13(2): 725-729.
- [Background] Jin Y, Chen J, Jiang Y, Yu B. Evaluation of a sexual abuse prevention education program for school-age children in China: a comparison of teachers and parents as instructors. Health Educ Res. 2017 Aug 1;32(4):364-373. doi: 10.1093/her/cyx047. PMID 28854573
- [Background] Huang S, Cui C. Preventing Child Sexual Abuse Using Picture Books: The Effect of Book Character and Message Framing. J Child Sex Abus. 2020 May-Jun;29(4):448-467. doi: 10.1080/10538712.2020.1719449. Epub 2020 Feb 28. PMID 32109197
- [Background] Czerwinski F, Finne E, Alfes J, Kolip P. Effectiveness of a school-based intervention to prevent child sexual abuse-Evaluation of the German IGEL program. Child Abuse Negl. 2018 Dec;86:109-122. doi: 10.1016/j.chiabu.2018.08.023. Epub 2018 Oct 1. PMID 30278285
- [Background] Manheim M, Felicetti R, Moloney G. Child Sexual Abuse Victimization Prevention Programs in Preschool and Kindergarten: Implications for Practice. J Child Sex Abus. 2019 Aug-Sep;28(6):745-757. doi: 10.1080/10538712.2019.1627687. Epub 2019 Jun 20. PMID 31219780
- [Background] Pulido ML, Dauber S, Tully BA, Hamilton P, Smith MJ, Freeman K. Knowledge Gains Following a Child Sexual Abuse Prevention Program Among Urban Students: A Cluster-Randomized Evaluation. Am J Public Health. 2015 Jul;105(7):1344-50. doi: 10.2105/AJPH.2015.302594. Epub 2015 May 14. PMID 25973809
- [Background] White C, Shanley DC, Zimmer-Gembeck MJ, Walsh K, Hawkins R, Lines K, Webb H. Promoting young children's interpersonal safety knowledge, intentions, confidence, and protective behavior skills: Outcomes of a randomized controlled trial. Child Abuse Negl. 2018 Aug;82:144-155. doi: 10.1016/j.chiabu.2018.05.024. Epub 2018 Jun 11. PMID 29902697
- [Background] Wurtele SK. Teaching young children personal body safety. The Body Safety Training Workbook. 2007. University of Colorado: Colorado Springs.
- [Background] Akgül E, Darak S, Sisman FN, Ergun A. Effect of the Nurse-Led. Journal of Psychiatric Nursing. 2021; 12(2): 156-164.
- [Background] Citak Tunc G, Gorak G, Ozyazicioglu N, Ak B, Isil O, Vural P. Preventing Child Sexual Abuse: Body Safety Training for Young Children in Turkey. J Child Sex Abus. 2018 May-Jun;27(4):347-364. doi: 10.1080/10538712.2018.1477001. Epub 2018 Jun 1. PMID 29856274
- [Background] Irmak TY, Kızıltepe R, Aksel Ş, Güngör D, Eslek D. Mika ile kendimi korumayı öğreniyorum: Cinsel istismarı önleme programının etkililiği ["I am learning to protect myself with Mika": The effectiveness of a sexual abuse prevention program]. Türk Psikoloji Dergisi. 2018; 33(81): 41-61.
- [Background] Warraitch A, Amin R, Rashid A. Evaluation of a school-based sexual abuse prevention program for female children with intellectual disabilities in rural Pakistan- A feasibility study. Appl Nurs Res. 2021 Feb;57:151391. doi: 10.1016/j.apnr.2020.151391. Epub 2020 Nov 25. PMID 33549294
- [Background] Bustamante G, Andrade MS, Mikesell C, Cullen C, Endara P, Burneo V, Yepez P, Avila Saavedra S, Ponce P, Grunauer M. "I have the right to feel safe": Evaluation of a school-based child sexual abuse prevention program in Ecuador. Child Abuse Negl. 2019 May;91:31-40. doi: 10.1016/j.chiabu.2019.02.009. Epub 2019 Feb 26. PMID 30822629
- [Background] Kim SJ, Kang KA. Effects of the Child Sexual Abuse Prevention Education (C-SAPE) Program on South Korean Fifth-Grade Students' Competence in Terms of Knowledge and Self-Protective Behaviors. J Sch Nurs. 2017 Apr;33(2):123-132. doi: 10.1177/1059840516664182. Epub 2016 Sep 20. PMID 27573418
- [Background] Jones C, Scholes L, Rolfe B, Stieler-Hunt C. A serious-game for child sexual abuse prevention: An evaluation of orbit. Child Abuse Negl. 2020 Sep;107:104569. doi: 10.1016/j.chiabu.2020.104569. Epub 2020 Jun 11. PMID 32535338
- [Background] Tutty LM. Child sexual abuse prevention programs: evaluating Who Do You Tell. Child Abuse Negl. 1997 Sep;21(9):869-81. doi: 10.1016/s0145-2134(97)00048-3. PMID 9298264
- [Background] Yılmaz Y, Cenkseven-Önder F. The Adaptation of Children's Knowledge of Abuse Questionnaire-Revised (CKAQ-R) to Turkish: Validity and reliability study. Elementary Education Online. 2020; 19(1): 384-392.
- See also: The California Evidence-Based Clearinghouse for Child Welfare. (CEBC). Prevention of Child Abuse and Neglect (Primary) Programs — https://www.cebc4cw.org/topic/prevention-of-child-abuse-and-neglect-primary-programs/